CLINICAL TRIAL: NCT01685320
Title: Force and Pressure Distribution Using Macintosh and GlideScope Laryngoscopes in Normal Airway: an in Vivo Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Massimiliano Carassiti, Professor, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PressureCara
Record Dates: First submitted 2012-09-07; First posted 2012-09-14 (Estimated); Results first posted 2013-03-13 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Tracheal Intubation; Laryngoscopy
Keywords: Force; Pressure; Intubation; laryngoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Direct laryngoscope (Active Comparator): Includes cases in which the forces applied by Macintosh direct laryngoscope onto soft tissue of the pharynx during glottis visualization and intubation were measured.
  Interventions: Procedure: Forces applied by laryngoscope
- Indirect laryngoscope (Active Comparator): Includes cases in which the forces applied by GlideScope indirect laryngoscope onto soft tissue of the pharynx during glottis visualization and intubation were measured.
  Interventions: Procedure: Forces applied by laryngoscope

INTERVENTIONS:
Procedure: Forces applied by laryngoscope — Force and pressure distribution applied by direct or indirect laryngoscope during glottis visualization and intubation were measured using film pressure transducers.

SUMMARY:
Forces applied on soft upper tissues by different laryngoscope blades during direct laryngoscopy and intubation are considered to be major stimuli to cause serious damages to the patients. The aim of this study is to compare the force and pressure applied to soft tissue in order to achieve the same glottis view comparing direct laryngoscopy and videolaryngoscopy in vivo.

DETAILED DESCRIPTION:
Forces applied on soft upper tissues by different laryngoscope blades during direct laryngoscopy and intubation are considered to be major stimuli to cause serious damages to the patients, such as local injures to incisors, larynx and spinal column, or hemodynamic changes in heart rate and/or blood pressure due to autonomic nervous system stimulation.

In order to reduce risk of such injures, indirect videolaryngoscopy provides the advantage of an easier laryngeal visualization with less need for the mouth-pharyngeal-laryngeal axes alignment, thereby reducing the detrimental effects above mentioned.

The aim of this study is to measure the minimal force exertion to achieve not only glottis view but also a successful intubation, comparing GlideScope and Macintosh laryngoscope, in patients with normal airway conditions. Furthermore, The investigators measured the following parameters: pressure distribution upon the blade; time required to visualize the glottis; time required to complete oro-tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as American Society of Anesthesiologists physical status (ASA-PS) class 1 or 2
* Patients whose intubation was associated with a Cormack-Lehane grade 1

Exclusion Criteria:

* younger than 18 yrs
* older than 65 yrs
* body-mass index (BMI) between 18 and 30
* predicted difficult intubation according to SIAARTI (Italian Society Anaesthesia, Analgesia, Resuscitation and Intensive Care)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Carassiti, Professor, Principal Investigator — Campus BioMedico
Locations (1):
- University Hospital Campus BioMedico, Rome, Italy

REFERENCES:
- [Result] Carassiti M, Zanzonico R, Cecchini S, Silvestri S, Cataldo R, Agro FE. Force and pressure distribution using Macintosh and GlideScope laryngoscopes in normal and difficult airways: a manikin study. Br J Anaesth. 2012 Jan;108(1):146-51. doi: 10.1093/bja/aer304. Epub 2011 Sep 28. PMID 21965048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of recruitment period: January-October 2011. Type of location: Dept. of Anaesthesia, University School of Medicine Campus Bio-Medico, Rome, Italy.
Pre-assignment Details: After written consent, thirty adult patients scheduled for elective surgery under general anaesthesia (age between 18 and 65 years, body-mass index between 18 and 30, classified as ASA-PS class 1 or 2), were included in this study. Subjects likely to be difficult to intubate, according to the SIAARTI Recommendations, were excluded.
Groups:
- Direct Laryngoscope: Includes cases in which the forces applied by McIntosh direct laryngoscope onto soft tissue of the pharynx during glottis visualization and intubation were measured using film pressure transducers.
- Indirect Laryngoscope: Includes cases in which the forces applied by GlideScope indirect laryngoscope onto soft tissue of the pharynx during glottis visualization and intubation were measured using film pressure transducers.
Period: Overall Study
Arm/Group | Direct Laryngoscope | Indirect Laryngoscope
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Laryngoscope | Indirect Laryngoscope | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (12) | 44 (11) | 42.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  Italy | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Force Applied and Pressure Distribution Upon the Blade of Laryngoscopes During Tracheal Intubation.
Description: The pressure distribution exerted upon the tissues by the blade was measured (in Newton)through pressure film transducers put on the blade of both direct and indirect laryngoscopes, in order to compare the two devices.
Time Frame: Force measurement is referred to an average of 45 seconds in patients scheduled to undergo elective surgery under general anaesthesia
Population: We have utilized our previous in vitro study on manikin (Carassiti et al. Br J Anaesth 2012; 108: 146-151) as basis for the calculus of sample size in this research, considering 95% confidence interval (2-sided), power of 80%, ratio of sample size (Group B/Group A) = 1.
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Direct Laryngoscope | Indirect Laryngoscope
Number analyzed (Participants) | 15 | 15
Newton
  Measurements during glottis visualization | 16 (6) | 10 (3)
  Measurements during intubation | 40 (14) | 8 (4)

2. Secondary Outcome: Time Required to Visualize the Glottis and Complete Oro-tracheal Intubation
Description: Since the time needed for laryngoscopy and intubation could represent one of the major contributors to the stress response during these procedures, times to achieve the glottis visualization and to perform the entire intubation were recorded.
Time Frame: On average 20 seconds
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Direct Laryngoscope | Indirect Laryngoscope
Number analyzed (Participants) | 15 | 15
seconds
  Time measured during glottis visualization | 13 (1) | 7 (1)
  Time measured during intubation | 22 (3) | 20 (1)

ADVERSE EVENTS:
Description: Serious and/or other non-serious adverse events were not collected/assessed
Arm/Group | Direct Laryngoscope | Indirect Laryngoscope
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
1. Patients studied were classified with "normal airways", while difficult intubations were not considered.
2. We excluded patients with CL grade 2 or greater.
3. We employed only the Macintosh size 3 blade to avoid additional variables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes